CLINICAL TRIAL: NCT01973413
Title: Diabetes Assistant (DiAs) Control-to-Range (CTR) Nocturnal Closed-Loop Camp Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Marc Breton, Co-Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 001-Stanford
Record Dates: First submitted 2013-10-24; First posted 2013-10-31 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Artificial Pancreas Project; Diabetes Mellitus, Type 1; Insulin pump therapy; Continuous Glucose Monitors (CGM); Juvenile-Onset Diabetes; Autoimmune Diabetes; Closed-to-Range; Diabetes Assistant (DiAs)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed-Loop Control with DiAs System (Experimental): Subjects will use the Diabetes Assistant (DiAs) and will wear a Tandem t:slim insulin pump and a Dexcom G4 Platinum sensor with active low and high sensor glucose alarms. Subjects will be remotely monitored throughout the night in real time.
  Interventions: Device: Diabetes Assistant (DiAs); Device: Tandem t:slim Insulin Pump; Device: Dexcom G4 Platinum sensor
- Control Group, Sensor-Augmented Pump Therapy (Placebo Comparator): Subjects will wear a Tandem t:slim insulin pump and a Dexcom G4 Platinum sensor with active low and high sensor glucose alarms. They will not use the Diabetes Assistant (DiAs) nor have remote monitoring.
  Interventions: Device: Tandem t:slim Insulin Pump; Device: Dexcom G4 Platinum sensor

INTERVENTIONS:
Device: Diabetes Assistant (DiAs) — The Control-to-Range (CTR) algorithm that will be used in DiAs will automatically adjusts insulin delivery in response to CGM values that have exceeded or are predicted to exceed the bounds of a pre-specified blood glucose range.
  Arms: Closed-Loop Control with DiAs System
Device: Tandem t:slim Insulin Pump — FDA, market-approved insulin pump.
Device: Dexcom G4 Platinum sensor — FDA, market-approved continuous glucose monitor (CGM)

SUMMARY:
The primary goal is to test the function of the Diabetes Assistant (DiAs) enhanced control-to-range (CTR) controller in a closely monitored diabetes camp setting. The camp setting will allow us to obtain pilot efficacy data.

DETAILED DESCRIPTION:
The first phase of this study will test the feasibility of initializing the DiAs CTR system in a clinical research center. We will test the procedures that will occur with the camp studies, from consenting the subjects, obtaining morning glucose readings, initializing the sensor in the early afternoon, having some light activity in the evening, a bedtime snack, and initializing the closed-loop system within 30 minutes before they go to bed. We will also test how the system performs using the same calibration and blood glucose monitoring that will be done at camp. In the inpatient study we will mimic some camp activities by having the subjects have 20-30 minutes of aerobic activity in the afternoon and in the evening after dinner. The data from the inpatient studies will be reviewed by the Data Safety Monitoring Board (DSMB) before we proceed with the Phase 2 summer camp studies.

The second phase of this proposal is the "in-camp" studies. The same health care providers that conducted the inpatient studies will be conducting the camp studies. They will be monitoring all campers on closed-loop control in real-time. Participants will be randomized to either closed-loop (experimental) or sensor-augmented therapy (control) for the first night and then crossed over every other night to the other therapy over the course of the 5- to 6-day camp session (i.e. on DiAs CTR every other night). Those assigned to DiAs CTR control will be remotely monitored throughout the night. Those assigned to the control group will not have remote monitoring overnight, but they will be wearing a Dexcom G4Platinum sensor with active low and high sensor glucose alarms. Initial studies will be done at a camp with older children and camp staff who are aged 15-35 years of age, with at least 5 subjects between 15 to 18 years old. If these studies are safe (after DSMB review) we will do additional camps and include children 10-14 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and a Medtronic, Animas or Tandem insulin infusion pump for at least 3 months
2. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide levels and antibody determinations are not required.
3. Age 10.0 - 35 years
4. Willingness to use a Sure-T or Contact Detach infusion set while at camp

Exclusion Criteria:

1. Diabetic ketoacidosis in the past month
2. Hypoglycemic seizure or loss of consciousness in the past 3 months
3. History of seizure disorder (except for hypoglycemic seizure)
4. Using an OmniPod insulin infusion pump
5. History of any heart disease including coronary artery disease, heart failure, or arrhythmias
6. Cystic fibrosis
7. Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
8. History of ongoing renal disease (other than microalbuminuria).
9. Insulin pump users who supplement with injected intermediate or long acting insulin.
10. Subjects who take other anti-diabetic medications other than insulin..
11. Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:
12. Inpatient psychiatric treatment in the past 6 months
13. Uncontrolled adrenal disorder
14. Abuse of alcohol
15. Pregnancy (verbal denial of pregnancy obtained with telephone informed consent, pregnancy test performed at camp before study devices are assigned).
16. Sexually active females who do not practice acceptable contraceptive methods to prevent pregnancy.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University; Marc Breton, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- Stanford University, Los Gatos, California, United States

REFERENCES:
- [Result] Ly TT, Breton MD, Keith-Hynes P, De Salvo D, Clinton P, Benassi K, Mize B, Chernavvsky D, Place J, Wilson DM, Kovatchev BP, Buckingham BA. Overnight glucose control with an automated, unified safety system in children and adolescents with type 1 diabetes at diabetes camp. Diabetes Care. 2014 Aug;37(8):2310-6. doi: 10.2337/dc14-0147. Epub 2014 May 30. PMID 24879841

RESULTS

PARTICIPANT FLOW:
Groups:
- Inpatient Study: The first phase of this study tested the feasibility of initializing the DiAs CTR system in a clinical research center. We tested the procedures that would occur with the camp studies, from consenting the subjects, obtaining morning glucose readings, initializing the sensor in the early afternoon, having some light activity in the evening, a bedtime snack, and initializing the closed-loop system within 30 minutes before they go to bed. We also tested how the system would perform using the same calibration and blood glucose monitoring that would be done at camp. In the inpatient study mimicked some camp activities by having the subjects have 20-30 minutes of aerobic activity in the afternoon and in the evening after dinner. The data from the inpatient studies was reviewed by the Data Safety Monitoring Board (DSMB) before we proceeded with the Phase 2 summer camp studies.
- Camp Study: The second phase of this proposal was the "in-camp" studies. The same health care providers that conducted the inpatient studies conducted the camp studies. They monitored all campers on closed-loop control in real-time. Participants were randomized to either closed-loop (experimental) or sensor-augmented therapy (control) for the first night and then crossed over every other night to the other therapy over the course of the 5- to 6-day camp session (i.e. on DiAs CTR every other night). Since participants were not always successfully completing a closed-loop control night, the pattern could not hold throughout the entire trial. Thus, there are numerous intervention sequences.
  Those assigned to DiAs closed-loop control were remotely monitored throughout the night. Those assigned to the control group were not monitored remotely overnight, but they were wearing Dexcom G4 Platinum sensors with active low and high sensor glucose alarms.
Period: Overall Study
Arm/Group | Inpatient Study | Camp Study
Started | 12 | 20
Completed | 11 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inpatient Study | Camp Study | Total
Number analyzed (Participants) | 12 | 20 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (2.1) | 15.3 (2.9) | 15.3 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 6 | 10 | 16
HbA1c [Mean (Standard Deviation); unit: percent of glycated hemoglobin] — Glycated hemoglobin, estimate of average blood glucose over past 3 months
  percent of glycated hemoglobin | 8.7 (0.7) | 8.1 (1.1) | 8.4 (1.0)
Diabetes Duration [Mean (Standard Deviation); unit: years] — Time since diagnosis of type 1 diabetes
  years | 7.6 (4.6) | 5.6 (3.5) | 6.4 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Time Near Normoglycemia
Description: Percent of time in a glucose target range of 70-150 mg/dl during camp study.
  Participants were randomized to either closed-loop (experimental) or sensor-augmented pump therapy (control) for the first night and then crossed over every other night to the other therapy over the course of the 5- to 6-day camp session. Thus there were ~60 nights of data for each intervention. However, data from closed-loop nights during which there were technical problems such as infusion set failure, sensor error >20%, or pump failure resulting in a >60-min interruption to closed-loop control were removed to allow for analysis of algorithm performance. Only nights with a minimum of 5 hours of closed-loop were included, and all glucose data were included in the analysis. For comparison, only data from nights during which sensor error was, <20% with a minimum of 5 hours were included in the control group.
Time Frame: 6 nights
Population: Data from OCL nights during which there were technical problems (infusion set failure, sensor error >20%, pump failure with >60-min interruption to closed-loop) were removed. Only nights with a minimum of 5h of OCL were included. For control, only data from nights where sensor error was <20% with a minimum of 5h were included.
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Total Nights of Data
Groups:
- Experimental: Closed-Loop Control: Subjects will use the Diabetes Assistant (DiAs) and will wear a Tandem t:slim insulin pump and a Dexcom G4 Platinum sensor with active low and high sensor glucose alarms. Subjects will be remotely monitored throughout the night in real time.
  Diabetes Assistant (DiAs): The Control-to-Range (CTR) algorithm that will be used in DiAs will automatically adjusts insulin delivery in response to CGM values that have exceeded or are predicted to exceed the bounds of a pre-specified blood glucose range.
- Control: Sensor-Augmented Pump Therapy: Subjects will wear a Tandem t:slim insulin pump and a Dexcom G4 Platinum sensor with active low and high sensor glucose alarms. They will not use the Diabetes Assistant (DiAs) nor have remote monitoring.
Arm/Group | Experimental: Closed-Loop Control | Control: Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 20 | 20
Number analyzed (Total Nights of Data) | 41 | 39
percentage of time | 73 [50 to 89] | 52 [24 to 83]
Statistical Analysis 1: Comparison: Experimental: Closed-Loop Control vs Control: Sensor-Augmented Pump Therapy; Test type: Non-Inferiority or Equivalence — Significance level of 0.05, 90% power, required 48 nights of OCL and 48 control nights to detect a 20% improvement; p = 0.037, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Overnight Glucose
Description: Mean overnight glucose during camp study.
  Participants were randomized to either closed-loop (experimental) or sensor-augmented pump therapy (control) for the first night and then crossed over every other night to the other therapy over the course of the 5- to 6-day camp session. Thus there were ~60 nights of data for each intervention. However, data from closed-loop nights during which there were technical problems such as infusion set failure, sensor error >20%, or pump failure resulting in a >60-min interruption to closed-loop control were removed to allow for analysis of algorithm performance. Only nights with a minimum of 5 hours of closed-loop were included, and all glucose data were included in the analysis. For comparison, only data from nights during which sensor error was, <20% with a minimum of 5 hours were included in the control group.
Time Frame: 6 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: Total Nights
Arm/Group | Experimental: Closed-Loop Control | Control: Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 20 | 20
Number analyzed (Total Nights) | 41 | 39
mg/dL | 140 (18) | 147 (36)
Statistical Analysis 1: Comparison: Experimental: Closed-Loop Control vs Control: Sensor-Augmented Pump Therapy; Test type: Superiority or Other; p = 0.340, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Glycemic Events
Description: Number of nights with >= 1 hypo- and hyperglycemic event occurring overnight during the camp study.
  Participants were randomized to either closed-loop (experimental) or sensor-augmented pump therapy (control) for the first night and then crossed over every other night to the other therapy over the course of the 5- to 6-day camp session. Thus there were ~60 nights of data for each intervention. However, data from closed-loop nights during which there were technical problems such as infusion set failure, sensor error >20%, or pump failure resulting in a >60-min interruption to closed-loop control were removed to allow for analysis of algorithm performance. Only nights with a minimum of 5 hours of closed-loop were included, and all glucose data were included in the analysis. For comparison, only data from nights during which sensor error was, <20% with a minimum of 5 hours were included in the control group.
Time Frame: 6 nights
Population: as for outcome 1
Measure: Number; unit: nights with >= 1 event
Units Other Than Participants: Total Number of Nights
Groups:
- Experimental: Closed-Loop Control: Subjects will use the Diabetes Assistant (DiAs) and will wear a Tandem t:slim insulin pump and a Dexcom G4 Platinum sensor with active low and high sensor glucose alarms. Subjects will be remotely monitored throughout the night in real time.
  Diabetes Assistant (DiAs): The Control-to-Range (CTR)algorithm that will be used in DiAs will automatically adjusts insulin delivery in response to CGM values that have exceeded or are predicted to exceed the bounds of a pre-specified blood glucose range.
Arm/Group | Experimental: Closed-Loop Control | Control: Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 20 | 20
Number analyzed (Total Number of Nights) | 41 | 39
nights with >= 1 event
  Hyperglycemic (>250mg/dl) | 4 | 4
  Hypoglycemic (<70mg/dl) | 7 | 14

ADVERSE EVENTS:
Arm/Group | Experimental: Closed-Loop Control | Control: Sensor-Augmented Pump Therapy
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/20
Other Adverse Events (participants affected / at risk) | 0/32 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No